CLINICAL TRIAL: NCT04822519
Title: RISK FACTORS OF GALL BLADDER STONE FORMATION
Brief Title: RISK FACTORS OF GALL BLADDER STONE
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Elbadry Elrabie, Resident in Tropical Medicine and Gastroenterology Department, Sohag University
Other Study IDs: Soh-Med-21-03-03
Record Dates: First submitted 2021-03-12; First posted 2021-03-30 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2021-03

CONDITIONS: Gall Stone
Keywords: Risk factors ,gallbladder stone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gallbladder disease is a significant health burden in the developed world and its prevalence has risen by more than 20% in the past three decades In the United States, 20-25 million individuals are affected by gallbladder disease, resulting in an average annual treatment cost of $6.2 billion Obesity, diet, rapid weight loss, metabolic syndrome, and conditions such as cirrhosis, Crohn's disease, irritable bowel syndrome, and gallbladder stasis increase the risk of gallstone formation Surgical removal of the gallbladder, cholecystectomy, is the most recommended treatment for gallbladder disease; however, the procedure increases the risk of non-alcoholic fatty liver disease, cirrhosis and metabolic effects

DETAILED DESCRIPTION:
Gallbladder disease is a significant health burden in the developed world and its prevalence has risen by more than 20% in the past three decades .

In the United States, 20-25 million individuals are affected by gallbladder disease, resulting in an average annual treatment cost of $6.2 billion Obesity, diet, rapid weight loss, metabolic syndrome, and conditions such as cirrhosis, Crohn's disease, irritable bowel syndrome, and gallbladder stasis increase the risk of gallstone formation .

Surgical removal of the gallbladder, cholecystectomy, is the most recommended treatment for gallbladder disease; however, the procedure increases the risk of non-alcoholic fatty liver disease, cirrhosis and metabolic effects .

Oral dissolution therapy using ursodeoxycholic acid is currently one of the leading non-invasive alternative treatments for gallstones. Ursodeoxycholic acid dissolves small cholesterol gallstones by decreasing hepatic secretion of cholesterol and lowering the chances of unsaturated gallbladder bile formation Although oral dissolution therapy has proven to be a safe alternative to cholecystectomy, it has a gallstone recurrence rate of 50%-70% at 12 years post-treatment .

The high incidence rate and treatment cost associated with gallbladder disease have encouraged the search for preventative strategies. In approximately 75% of cases, impaired gallbladder motility results from the accumulation of cholesterol gallstones. Therefore, agents that reduce lipid concentrations or improve gallbladder motility may reduce the need for surgical interventions and/or the use of potentially harmful pharmaceutical products .

ELIGIBILITY:
Inclusion Criteria:

Adult patients who have gall bladder stone(s)

Exclusion Criteria:

Child -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include all adult patients with gallstones admitted to Tropical Medicine Department, Sohage University Hospital.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to unravel the mechanisms responsible for the increased risk of gall stone disease. | 15 weeks
  All patients will be subjected to:-
  Complete history taking:
  With stress on:-
  * Age sex ( female or male ) comorbid condition (diabetes or hypersensitive).
  * History of taking lipid lowering drugs.
  Thorough clinical examination:
  General examination vital sign ( pulse / blood pressure) height ( centimetre) weight ( kilogram ) body mass index( kg / m2) . Abdominal examination ( organomegly / percussion ).
  Laboratory Investigation:
  1. Lipid profile (total cholesterol, triglyceride, HDL, LDL, VLDL(
  2. Abdominal ultrasound.
  3. Thyroid function test.(T3 / T4)
  4. Estrogen.
  5. Random blood suger

CONTACTS AND LOCATIONS:
Locations (1):
- at the department of tropical medicine and gastroenterology at sohag University Hospital., Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Undecided